CLINICAL TRIAL: NCT05775263
Title: Validation of UK Protocols to Exclude Brain Blood Flow During Normothermic Regional Perfusion (NRP)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: PO3027
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Cerebral Blood Flow

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A-NRP
  Interventions: Procedure: CT angiogram
- TA-NRP
  Interventions: Procedure: CT angiogram

INTERVENTIONS:
Procedure: CT angiogram — CT angiography of the brain 30 minutes from establishment of NRP

SUMMARY:
This study aims to evaluate both Abdominal Normothermic Regional Perfusion (A-NRP) and Thoracoabdominal-NRP (TA-NRP) techniques, proving that brain blood flow is not resumed during NRP. This will be assessed through the use of two modalities: CT angiogram of the brain and continuous Hb02 readings. The study group hypothesise that such assessment methods will provide evidence to indicate that brain blood flow is not present during NRP and promote trust in the use of such novel techniques in routine practice.

ELIGIBILITY:
Inclusion Criteria:

* DCD donors in Cambridge University Hospital
* Planned A-NRP
* Consent for study has been obtained
* Those who meet the appropriate criteria for DCD donation following WOLST
* ≥ 18 years of age
* ≤ 75 years of age

Exclusion Criteria:

* DBD organ donors
* DCD organ donations outside of Cambridge University Hospital
* DCD donors without planned A-NRP
* DCD donors whose family have withheld consent for brain blood flow investigations.
* Patients who do not meet the appropriate criteria for DCD donation following WOLST
* Patients with injuries that will physically prevent use of the necessary assessment methods

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Donation after Circulatory Death (DCD) organ donors
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
CT angiogram | 30 minutes from establishment of NRP
  Brain blood flow

SECONDARY OUTCOMES:
Cerebral oximetry | Prior to withdrawal of life sustaining treatment to 30 minutes after establishment of NRP
  HbO2 measurements (O2Hbi (Delta oxygenated), HHbi (Delta deoxygenated), and cHbi (Delta total))